CLINICAL TRIAL: NCT00295971
Title: Stem Cell Enriched, T Cell Depleted Haplocompatible Peripheral Blood Transplantation for Children With Myelodysplastic Disease, Leukemia, Marrow Failure Syndromes, or Severe Immunodeficiency Diseases
Brief Title: Donor Stem Cell Transplant in Treating Young Patients With Myelodysplastic Syndrome, Leukemia, Bone Marrow Failure Syndrome, or Severe Immunodeficiency Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Morton Cowan, Professor, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000462168; UCSF-01151; UCSF-H411-17122-07
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Congenital Amegakaryocytic Thrombocytopenia; Leukemia; Myelodysplastic Syndromes; Severe Congenital Neutropenia
Keywords: childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; secondary acute myeloid leukemia; juvenile myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; severe congenital neutropenia; congenital amegakaryocytic thrombocytopenia; childhood chronic myelogenous leukemia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Congenital amegakaryocytic thrombocytopenia; Leukemia; Myelodysplastic Syndromes; Neutropenia, Severe Congenital, Autosomal Recessive 3; Leukemia, Myelomonocytic, Juvenile; Leukemia, Myeloid, Chronic-Phase; Anemia, Refractory, with Excess of Blasts | interventions — Antilymphocyte Serum; fludarabine phosphate; Thiotepa; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm of transplant (Experimental): Receiving haplocompatible T cell depleted peripheral blood stem cell transplant
  Interventions: Biological: anti-thymocyte globulin; Biological: therapeutic allogeneic lymphocytes; Drug: fludarabine phosphate; Drug: thiotepa; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: in vitro-treated peripheral blood stem cell transplantation; Radiation: total-body irradiation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: therapeutic allogeneic lymphocytes
Drug: fludarabine phosphate
Drug: thiotepa
Procedure: allogeneic bone marrow transplantation
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: in vitro-treated peripheral blood stem cell transplantation
Radiation: total-body irradiation

SUMMARY:
RATIONALE: Giving chemotherapy and total body irradiation before a donor bone marrow transplant or peripheral blood stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving antithymocyte globulin and removing the T cells from the donor cells before transplant may stop this from happening.

PURPOSE: This phase I trial is studying the side effects and best dose of donor T cells and antithymocyte globulin when given together with chemotherapy and total-body irradiation in treating young patients who are undergoing T-cell depleted donor stem cell transplant for myelodysplastic syndrome, leukemia, bone marrow failure syndrome, or severe immunodeficiency disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy and toxicity of stem cell-enriched, T-cell-depleted, haplocompatible allogeneic hematopoietic stem cell transplantation in children with high-risk myelodysplastic syndromes, high-risk leukemia, severe acquired or congenital cytopenias, or primary immunodeficiency diseases.
* Determine the toxicity of a fludarabine and thiotepa-containing regimen in combination with lower doses of antithymocyte globulin in these patients.
* Determine the engraftment rate in patients treated with this regimen.
* Define T-cell reconstitution in these patients.
* Determine the toxicity and effects of administering stem cell and T-cell boosts after transplantation on hematopoiesis and immune reconstitution in these patients.

OUTLINE: This is a dose-escalation study of donor CD3+ cells and antithymocyte globulin (ATG).

* Cytoreductive regimen: Patients undergo total body irradiation twice daily on days -9 to -7. Patients also receive fludarabine IV on days -6 to -2, thiotepa IV every 12 hours on day -6, and ATG IV on days -5 to -2.
* Transplantation: Patients undergo CD34-enriched, T-cell-depleted, haplocompatible allogeneic peripheral blood stem cell or bone marrow transplantation on day 0.
* Donor T-cell infusion:Patients with no active graft-vs-host disease and evidence of engraftment but low absolute CD34+ lymphocyte count at 12 weeks post transplant may receive donor CD3+ cells at 4-week intervals.
* Donor stem cell boost: Patients with engraftment but either cytokine or transfusion dependent at 12 weeks post transplant may receive a boost of donor CD34+ cells.

Cohorts of 3-6 patients receive escalating doses of donor CD3+ cells and ATG until the optimum is determined. The optimum dose is defined as the dose at which both engraftment and T-cell recovery occur, without dose-limiting toxicity, in ≥ 5 of 6 patients.

After the completion of study treatment, patients are followed periodically for 5 years and then every 5 years thereafter.

PROJECTED ACCRUAL: A total of 21 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following:

  * Acute lymphoblastic leukemia in ≥ 2nd remission or delayed remission induction
  * High-risk myelodysplastic syndromes

    * Refractory anemia with excess blasts (RAEB)
    * RAEB in transformation
  * Chronic myelogenous leukemia in second chronic phase

    * No accelerated phase (> 5% blasts in marrow)
  * Juvenile myelomonocytic leukemia
  * Acute nonlymphoblastic leukemia in > 1st remission or induction failure and < 30% blasts in marrow
  * Severe aplastic anemia, defined as absolute neutrophil count < 500/mm^3 and platelet and/or red blood cell transfusion dependent

    * Unresponsive to immunosuppressive therapy
    * No Fanconi's anemia
  * Congenital marrow aplasias unresponsive to cytokines and transfusion dependent
  * Inherited immunodeficiency disease involving neutrophils or lymphocytes, including any of the following:

    * Chediak-Higashi disease
    * Wiskott-Aldrich syndrome
    * Combined immunodeficiency disease (Nezelof's)
    * Hyper IgM syndrome
* No relapsed disease
* Haplocompatible related donor, including parent, cousin, aunt, uncle, grandparent, half-sibling, or sibling (≥ 12 years of age), available

  * 2 or 3 HLA antigen mismatch
  * At least a 3 HLA antigen genotypic match
  * No closely matched related or unrelated donor available in sufficient time to do the transplant

PATIENT CHARACTERISTICS:

* No active hepatitis or cytomegalovirus infection
* Cardiac ejection fraction ≥ 30%
* Creatinine clearance ≥ 70 mL/min
* DLCO ≥ 70% of predicted
* No active infection
* No HIV positivity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2005-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Engraftment at 4 weeks post bone marrow transplantation through 100 days | 100 days

SECONDARY OUTCOMES:
Survival assessed monthly for 6 months, every 3 months for 2 years, every 6 months for 1 year, and then yearly for 5 years post transplantation | 1 year
Disease-free survival and infection assessed monthly for 6 months, every 3 months for 2 years, every 6 months for 1 year, and then yearly for 5 years post transplantation | 1 year
Graft-versus-host disease assessed monthly for 6 months, every 3 months for 2 years, every 6 months for 1 year, and then yearly for 5 years post transplantation | 2 years
CD4 count in blood < 100/mm³ at 12 weeks | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Morton J. Cowan, MD, Study Chair — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina